CLINICAL TRIAL: NCT04378140
Title: Retention and Durability of the Anterior Zirconia Wing Bridge
Status: Active, not recruiting | Type: Observational
Sponsor: Roseman University of Health Sciences (Other)
Responsible Party: Principal Investigator, David McMillan, Principal Investigator, Roseman University of Health Sciences
Other Study IDs: 1164902
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Missing Teeth; Partial-edentulism
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: zirconia wing bridge — The zirconia wing bridge consists of an artificial tooth made out of zirconia and porcelain on the front side with two zirconia wings that are bonded (glued) onto the back of the two adjacent teeth in the patient's mouth.

SUMMARY:
This study is a clinical trial to determine the retention and durability of the anterior zirconia wing bridge. The type of zirconia-wing bridge the investigators are researching in this study has two wings which generally have three countersunk holes (meaning that the circumference of the outer portion of the hole is larger than the inner part of the hole). Composite resin (dental filling material) is placed in the holes as well as under and around the wings.

Twelve patients will have bridges placed and be evaluated every 6 months (ideally) to determine if the bridge is staying in place (retention) and if it is resistant to fracture (durability).

DETAILED DESCRIPTION:
For patients missing an anterior tooth, the treatment options available include a dental implant, a removable partial denture, or a bridge. Some patients may not desire an implant due to the surgical nature, the limited bone available or the high cost. Removable partial dentures are relatively inexpensive but are undesirable for many patients due to the limited esthetics, trouble speaking and annoyance of an oral prosthesis. Traditional bridges use adjacent teeth as abutments and replace the missing tooth. However, these require the removal of 1-2 mm of tooth structure on adjacent teeth provide room for the porcelain of the bridge.

Decades ago, the option for a conservative bridge was primarily found in the Maryland bridge, which had two metal wings that were cemented or bonded on to two abutments. Though conservative, the Maryland Bridge did not enjoy a high reputation because of the high rate of debonding (falling off).

In the last several decades, the use of zirconia as a restorative material in dentistry has dramatically risen due to its toughness, resemblance in color to natural teeth, and affordability. Also, composite resin bonding agents (adhesive for dental fillings) have increased in strength and effectiveness. With these two advancements, the possibility of overcoming the some of the previous shortcomings with the Maryland Bridge is more of a reality.

The type of zirconia-wing bridge we are researching in this study has two wings which generally have three countersunk holes (meaning that the circumference of the outer portion of the hole is larger than the inner part of the hole). Composite resin (dental filling material) is placed in the holes as well as under and around the wings.

In summary, the zirconia-wing bridge presents a desirable alternative to traditional options for missing anterior teeth. With the advancements in resin-bonding and zirconia, this study seeks to examine how these combined elements can be used in the zirconia-wing bridge to maximize durability and retention in clinical scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Registered patient at Roseman University of Health Sciences in South Jordan, Utah who has undergone a health and dental screening
* One missing anterior tooth
* Adjacent teeth to the missing tooth must be non-restored or minimally-restored in with gums that have pockets of 4 millimeters or less
* Fluent in English or Spanish

Exclusion Criteria:

* Patients who are not registered at Roseman University of Health Sciences in South Jordan, Utah
* Patients who are unable to attend 6-month recall appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of both genders, ages 18 and above with one missing anterior teeth that has periodontal pockets of no more than 4 mm with abutment teeth being non-restored or minimally restored.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2030-12-20 (Estimated); Study Completion 2030-12-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants with bridges still bonded to the teeth (retention) | 2 years observation
  Determines how long the bridge stays bonded to the patient's teeth

SECONDARY OUTCOMES:
Number of participants with bridges that have no fractures (durability) | 2 years observation
  Determine if there is any fracturing of the zirconia

CONTACTS AND LOCATIONS:
Overall Officials: David G McMillan, DDS, Principal Investigator — Roseman University of Health Sciences
Locations (1):
- Roseman University of Health Sciences, South Jordan, Utah, United States

DOCUMENTS (1):
  • Informed Consent Form (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT04378140/ICF_000.pdf